CLINICAL TRIAL: NCT00540982
Title: Pilot Pharmacokinetic Study of Dose Adjustment of Vinorelbine in Patients With Varying Degree of Liver Dysfunction
Brief Title: Vinorelbine in Treating Patients With Advanced Solid Tumors That Have Not Responded to Treatment and Liver Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96032; P30CA033572 (NIH); CHNMC-96032; CDR0000567457 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Indocyanine Green; Lidocaine; Vinorelbine; Chromatography, High Pressure Liquid; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal Liver Function (Experimental)
  Interventions: Drug: indocyanine green; Drug: lidocaine; Drug: vinorelbine ditartrate; Other: high performance liquid chromatography; Other: intracellular fluorescence polarization analysis; Other: liquid chromatography; Other: mass spectrometry; Other: pharmacological study
- Mild Liver Dysfunction (Experimental)
  Interventions: Drug: indocyanine green; Drug: lidocaine; Drug: vinorelbine ditartrate; Other: high performance liquid chromatography; Other: intracellular fluorescence polarization analysis; Other: liquid chromatography; Other: mass spectrometry; Other: pharmacological study
- Moderate Liver Dysfunction (Experimental)
  Interventions: Drug: indocyanine green; Drug: lidocaine; Drug: vinorelbine ditartrate; Other: high performance liquid chromatography; Other: intracellular fluorescence polarization analysis; Other: liquid chromatography; Other: mass spectrometry; Other: pharmacological study
- Severe Liver Dysfunction (Experimental)
  Interventions: Drug: indocyanine green; Drug: lidocaine; Drug: vinorelbine ditartrate; Other: high performance liquid chromatography; Other: intracellular fluorescence polarization analysis; Other: liquid chromatography; Other: mass spectrometry; Other: pharmacological study

INTERVENTIONS:
Drug: indocyanine green — 0.5 mg/kg will be administered by IV push to determine clearance
Drug: lidocaine — 1 mg/kg will be administered to determine metabolic capacity
Drug: vinorelbine ditartrate — Varying doses ranging from 30 mg/m2 to 7.5 mg/m2 will be administered based upon liver function
Other: high performance liquid chromatography — Used to determine plasma concentrations of vinorelbine
Other: intracellular fluorescence polarization analysis — Used to determine concentration of lidocaine metabolic capacity
Other: liquid chromatography — Used to determine concentrations of vinorelbine and its metabolites
Other: mass spectrometry — Used to determine concentrations of vinorelbine and its metabolites
Other: pharmacological study — Determination of concentrations of vinorelbine and its metabolites

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This pilot trial is studying the side effects and best dose of vinorelbine in treating patients with advanced solid tumors that have not responded to treatment and liver dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES:

* To correlate indocyanine green and lidocaine metabolism with vinorelbine ditartrate pharmacokinetics in patients with advanced, refractory solid tumors and varying degrees of liver dysfunction.
* To determine the pharmacokinetics of vinorelbine ditartrate in these patients.
* To test a plan of dose adjustment for vinorelbine ditartrate administration in these patients.

OUTLINE: Patients are stratified according to extent of clinical liver dysfunction (normal vs mild vs moderate vs severe).

Patients receive dose-adjusted vinorelbine ditartrate IV over 10 minutes once weekly in the absence of disease progression or unacceptable toxicity. Patients achieving an objective complete response receive 2 additional courses of study therapy.

Patients undergo blood sample collection periodically during study for pharmacokinetic and pharmacodynamic correlative studies. Blood is also collected after patients receive lidocaine IV push and indocyanine green (ICG) IV push. Samples are analyzed for whole blood and plasma concentrations of vinorelbine ditartrate and its metabolites by high performance liquid chromatography (15) or by liquid chromatography/tandem mass spectrometry assay. Samples are also analyzed for ICG clearance and lidocaine hydrochloride metabolic capacity by fluorescent polarization immunoassay.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor

  * Any histology allowed
* Refractory to standard therapy OR no standard therapy exists

  * Previously untreated non-small cell lung cancer allowed, provided abnormal liver function is present, defined as moderate (group 3) or severe (group 4)
* Measurable disease not required

  * Present measurable disease requires baseline measurements within 4 weeks of study entry
* Patients with acute hepatitis from viral or drug etiologies should recover to a stable baseline prior to study therapy
* History of brain metastasis allowed, provided the following criteria are met:

  * Metastasis has been controlled by radiotherapy or surgery
  * Patient is not currently on corticosteroids
  * Neurologic status is stable

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 2 months
* ANC = 1,500/mm³
* Platelet count = 100,000/mm³
* Hemoglobin = 10 g/dL (transfusion to this level allowed)
* Creatinine < 1.5 mg/dL OR creatinine clearance > 60 mL/ min
* Patients with EKG evidence of first- or second-degree AV block or left or right bundle branch block are ineligible for the lidocaine bolus, but may otherwise be treated on this protocol
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent illness (e.g., cardiovascular, pulmonary, or central nervous system) that is poorly controlled or of such severity that the investigator deems unwise to enter the patient on protocol
* Must have ability to comply with study treatment and required tests
* Obstructive jaundice requires a drainage procedure prior to study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea therapy)
* No prior radiotherapy to > 30% of the bone marrow or more than standard adjuvant pelvic radiotherapy for rectal cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 1997-02-20 (Actual); Primary Completion 2010-05-20 (Actual); Study Completion 2010-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chao, Study Chair — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients with treatment-refractory solid tumors enrolled on the study.
Period: Overall Study
Arm/Group | All Patients
Started | 47
Normal Liver Function | 11
Mild Liver Dysfunction | 6
Moderate Liver Dysfunction | 18
Severe Liver Dysfunction | 12
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23
  Hispanic | 13
  Asian | 9
  African American | 2
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve
Description: Pharmacokinetics were evaluated in patients with sufficient dosing information and plasma concentration versus time data over 0-24 hours following vinorelbine infusion to allow calculation of area-under-the-curve from zero to 24 hours after infusion (AUC0-24). Furthermore, dose-normalization of AUC0-24 to the standard 30 mg/m2 dose was performed to allow evaluation of the relationship between liver function and AUC of vinorelbine. Data were collected at 0 and 24 hours post-dose.
Time Frame: 2 months post treatment
Population: Vinorelbine plasma AUC0-24 data were available for a total of 30 subjects.
Measure: Median (Full Range); unit: ng/ml x hr
Groups:
- Normal: Patients were administered weekly 30mg/m2 of vinorelbine as a short IV infusion (over 10 minutes maximum).
  Normal liver function was defined as bilirubin <1.5 mg/dL
- Mild: Patients were administered weekly 30mg/m2, 20mg/m2 or 15mg/m2 of vinorelbine as a short IV infusion (over 10 minutes maximum).
  Mild liver dysfunction defined as bilirubin <1.5 mg/dL and ≥1 of the following: AST/ALT 1.5-2.5 X ULN or ALK 1.5-3 X ULN
- Moderate: Patients were administered weekly 30mg/m2 or 15mg/m2 of vinorelbine as a short IV infusion (over 10 minutes maximum).
  Moderate liver dysfunction was defined as bilirubin 1.5-3.0 mg/dL and/or ≥1 of the following: AST/ALT >2.5 X ULN or ALK >3 X ULN.
- Severe: Patients were administered weekly 20mg/m2 or 7.5mg/m2 of vinorelbine as a short IV infusion (over 10 minutes maximum).
  Severe liver dysfunction was defined as bilirubin >3.0 mg/dL.
Arm/Group | Normal | Mild | Moderate | Severe
Number analyzed (Participants) | 10 | 4 | 12 | 4
ng/ml x hr | 271 [111 to 593] | 537 [366 to 812] | 341 [251 to 1318] | 324 [167 to 1090]

2. Primary Outcome: Number of Participants With Grade 3 and 4 Toxicities
Description: Grade 3 & 4 toxicities at least possible related to study drugs during any cycle of treatment. Toxicity graded according to Common Terminology Criteria for Adverse Events version 2.0.
Time Frame: 3 weeks after the stop of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Normal (30mg/m2): Normal Liver Function Group with 30 mg/m2 of Vinorelbine.
- Mild (30mg/m2): Mild Liver Dysfunction Group with 30 mg/m2 of Vinorelbine.
- Mild (20mg/m2): Mild Liver Dysfunction Group with 20 mg/m2 of Vinorelbine.
- Mild (15mg/m2): Mild Liver Dysfunction Group with 15 mg/m2 of Vinorelbine.
- Moderate (30mg/m2): Moderate Liver Dysfunction Group with 30 mg/m2 of Vinorelbine.
- Moderate (15mg/m2): Moderate Liver Dysfunction Group with 15 mg/m2 of Vinorelbine.
- Severe (20mg/m2): Severe Liver Dysfunction Group with 20 mg/m2 of Vinorelbine.
- Severe (7.5mg/m2): Severe Liver Dysfunction Group with 7.5 mg/m2 of Vinorelbine.
Arm/Group | Normal (30mg/m2) | Mild (30mg/m2) | Mild (20mg/m2) | Mild (15mg/m2) | Moderate (30mg/m2) | Moderate (15mg/m2) | Severe (20mg/m2) | Severe (7.5mg/m2)
Number analyzed (Participants) | 11 | 1 | 3 | 2 | 8 | 10 | 7 | 5
Participants
  Anemia | 1 | 0 | 2 | 0 | 1 | 3 | 1 | 0
  Lymphopenia | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Neutropenia | 4 | 1 | 2 | 1 | 7 | 4 | 4 | 0
  Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  Anorexia/weight loss | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Ascites | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cerebrovascular ischemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Confusion | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Constipation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Dehydration | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Diarrhea | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspnea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Edema | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Fatigue | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Generalized weakness | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Hallucinations | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypotension | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Hypertension | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infection (including febrile neutropenia) | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0
  Thromboembolism | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Abnormal LFTs | 0 | 1 | 0 | 0 | 1 | 3 | 3 | 3
  Hypercalcemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hyperglycemia | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 2
  Hyperkalemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypophosphatemia | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Neuropathy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Pain | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Petechiae/purpura | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Pulmonary hemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Elevated INR | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypokalemia | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0
  Hyponatremia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and graded throughout the study and until 30 days following the last dose of vinorelbine.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Normal (30mg/m2) | Mild (30mg/m2) | Mild (20mg/m2) | Mild (15mg/m2) | Moderate (30mg/m2) | Moderate (15mg/m2) | Severe (20mg/m2) | Severe (7.5mg/m2)
All-Cause Mortality (participants affected / at risk) | 11/11 | 1/1 | 3/3 | 2/2 | 8/8 | 10/10 | 7/7 | 5/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/1 | 0/3 | 0/2 | 3/8 | 0/10 | 4/7 | 0/5
Other Adverse Events (participants affected / at risk) | 11/11 | 1/1 | 3/3 | 2/2 | 7/8 | 10/10 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal (30mg/m2) (N=11) | Mild (30mg/m2) (N=1) | Mild (20mg/m2) (N=3) | Mild (15mg/m2) (N=2) | Moderate (30mg/m2) (N=8) | Moderate (15mg/m2) (N=10) | Severe (20mg/m2) (N=7) | Severe (7.5mg/m2) (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
(Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal (30mg/m2) (N=11) | Mild (30mg/m2) (N=1) | Mild (20mg/m2) (N=3) | Mild (15mg/m2) (N=2) | Moderate (30mg/m2) (N=8) | Moderate (15mg/m2) (N=10) | Severe (20mg/m2) (N=7) | Severe (7.5mg/m2) (N=5)
Cerebellar (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clinical (Physical Exam) (General disorders) | 4 (15) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (12) | 0 (0) | 3 (32)
Dysrhythmias (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid Retention (General disorders) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 3 (22)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage (General disorders) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 3 (22)
Infection (Infections and infestations) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (13) | 0 (0) | 3 (22)
Ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other Misc (General disorders) | 4 (35) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (19) | 0 (0) | 3 (39)
Pericardial (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 3 (22)
Stomatitis (Skin and subcutaneous tissue disorders) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 3 (22)
Weight (Food Intake) (Metabolism and nutrition disorders) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 3 (22)
Clinical Coagulation (Blood and lymphatic system disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (12) | 1 (1) | 3 (33) | 1 (1) | 5 (6) | 6 (44) | 7 (9) | 2 (10)
Lymphatics (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EF/CHF (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (2) | 3 (3) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (10) | 3 (3) | 2 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (19) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (8) | 0 (0) | 4 (17)
Diarrhea (Gastrointestinal disorders) | 5 (19) | 0 (0) | 1 (5) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 4 (14)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (19) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (10) | 1 (1) | 4 (16)
Vomiting (Gastrointestinal disorders) | 6 (19) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (7) | 0 (0) | 4 (16)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Edema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (17) | 1 (2) | 3 (13) | 2 (2) | 6 (7) | 9 (14) | 6 (7) | 5 (24)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 1 (1)
Fever (no infection) (General disorders) | 4 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 3 (20)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Oedema NOS (General disorders) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 0 (0) | 5 (12) | 1 (1) | 2 (8)
Pain (General disorders) | 4 (7) | 1 (2) | 1 (9) | 0 (0) | 4 (5) | 3 (10) | 3 (4) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Allergy (Immune system disorders) | 5 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 3 (22)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
(Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AGC (Investigations) | 5 (21) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (13) | 0 (0) | 3 (29)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (6) | 1 (2) | 1 (1) | 1 (1) | 5 (6) | 5 (20) | 6 (8) | 2 (9)
Alkaline Phosphatase (Investigations) | 4 (15) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (12) | 0 (0) | 3 (32)
Alkaline phosphatase increased (Investigations) | 4 (7) | 1 (2) | 3 (33) | 1 (1) | 6 (8) | 6 (44) | 5 (7) | 2 (10)
Amylase (Investigations) | 3 (9) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (6) | 0 (0) | 3 (19)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 1 (2) | 3 (33) | 1 (1) | 6 (8) | 6 (33) | 6 (8) | 2 (11)
Bilirubin (Investigations) | 4 (15) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (12) | 0 (0) | 3 (32)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 0 (0)
Creatinine (Investigations) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Fibrinogen (Investigations) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HGB/HCT (Investigations) | 5 (23) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (13) | 0 (0) | 3 (29)
Hyperbilirubinemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (8) | 1 (1) | 2 (10)
Hypercholesterolemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 4 (6) | 0 (0)
Leukopenia (Investigations) | 3 (4) | 0 (0) | 3 (16) | 0 (0) | 1 (2) | 4 (11) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Lymphopenia (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (8) | 1 (2) | 2 (7) | 0 (0) | 6 (8) | 2 (5) | 5 (6) | 0 (0)
Partial Thromboplastin Time (Investigations) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (3) | 4 (4) | 1 (3)
Platelets (Investigations) | 5 (23) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (13) | 0 (0) | 3 (29)
Prothrombin Time (Investigations) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
SGOT/SGT (Investigations) | 4 (15) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (12) | 0 (0) | 3 (32)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
WBC (Investigations) | 5 (23) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (13) | 0 (0) | 3 (29)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (6)
Weight loss (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 3 (24) | 1 (1) | 5 (5) | 2 (8) | 3 (3) | 1 (1)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (7) | 1 (2) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 1 (3) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (13) | 0 (0) | 3 (19)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (14) | 0 (0) | 2 (25) | 2 (3) | 0 (0) | 7 (22) | 0 (0) | 4 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 3 (8) | 1 (1) | 0 (0) | 6 (39) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (12) | 0 (0) | 1 (2) | 2 (3) | 1 (2) | 5 (17) | 2 (2) | 5 (23)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 3 (9) | 0 (0) | 3 (19)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 3 (8) | 2 (3) | 3 (19)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (4) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 5 (6) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cortical/State of Consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor Activity (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Nervous System Sensory (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (22) | 0 (0) | 1 (1) | 3 (10) | 0 (0) | 0 (0)
Mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (9) | 4 (5) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (27) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 5 (14) | 0 (0) | 3 (22)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Local Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes